CLINICAL TRIAL: NCT02551445
Title: A fMRI Pilot Study of the Effects of Cognitive Behavioural Therapy (Meal-support) in Eating Disorders.
Brief Title: A fMRI Pilot Study of the Effects of Meal-support in Eating Disorders.
Acronym: ET4AN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIEF-2011-299232
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gradual exposure to food stimuli (Experimental): The intervention entails 2 sessions of psychoeducation and a clinical assessment including a discussion on learned food-related fears, role of food-related fears in the maintenance of anorexia nervosa, anxiety and its time course, avoidance, exposure and habituation, irrational fears and safety behaviors; and 8 sessions of in vivo exposure to foods, starting from the least scary food of a hierarchy of threatening foods created by each patient. Each session will involve exposure to a new food item and patients will be encouraged to confront their fear by looking at and touching the chosen food item. They will also be encouraged to eat the food and reflect on the consequences of eating and assessing those relative to their fears (e.g. checking whether they have lost control or changed shape after eating).
  Interventions: Behavioral: Gradual exposure to food stimuli

INTERVENTIONS:
Behavioral: Gradual exposure to food stimuli — Patients with anorexia nervosa will be encouraged to confront their fears and avoidance in relation to food and will be gradually exposed to different food items during the sessions.

SUMMARY:
This study involves people with eating disorders and healthy volunteers (people who have never experienced an eating disorder). Participants are interviewed about their psychological and physical health by the experimenter and they have a simulated scan session (about 1 hour). Approximately 1 week after they attend the first study session. They are asked to complete questionnaires and computerized tasks (about 30 minutes) followed by the active scan (1 hour). During the brain scan they look at pictures and answer questions about the pictures. After the first study session, people with eating disorders receive an intensive meal-support intervention (in the following 3 months) aimed at reducing anxiety and fears related to food (10 sessions lasting about 60 min.). Three months after the first brain scan, participants with eating disorders and healthy controls receive a second assessment and brain scan. We hypothesized that the meal support intervention will be effective in: 1) targeting eating disorder symptoms (body mass index - BMI, primarily) and 2) producing functional changes in brain regions that underline food-related anxiety and avoidance.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is characterized by severe malnutrition. Patients report aversive experiences of re-feeding and frequently drop-out from treatment. This study will test the hypothesis that gradual and guided exposure to food is associated with increased body mass index (BMI) and reduced eating disorder psychopathology in patients with AN. It is also hypothesized that the intervention will lead to changes in brain activation in regions implicated in anticipatory anxiety and fear of food and emotion regulation (i.e. amygdala, insula, dorso-lateral prefrontal cortex [DLPFC]). Sixteen women with anorexia nervosa not receiving any interventions at the time of the study will be recruited from the community. Patients will complete a range of self-report measures and will undergo a functional magnetic resonance imaging (fMRI) scan before and after receiving 10 exposure therapy sessions over 3 months. A matched healthy control group (n=20) will also have two brain scans 3 months apart.

To be eligible for the study, participants will have to be female, proficient in English, right-handed, between 19 and 60 years. Participants in the clinical group will have to meet the DSM-IV-TR diagnostic criteria for anorexia nervosa. Participants in the healthy control group will be required to have a BMI between 18.5 and 25 kg/m² and no history of, or current, mood and anxiety disorders. Additional exclusion criteria will be: history of head trauma, hearing or visual impairment, neurological disease, claustrophobia, pregnancy, metal in the body which cannot be removed, history of (or current) drugs and/or alcohol abuse; acute suicidality, psychotropic medication (other than antidepressants in the patient group).

Pre- and post-intervention changes in patients' BMI, anxiety, eating disorders symptoms, mood and motivation to change will be assessed. Changes in brain activations in selected regions of interest, including the DLPFC, amygdala and insula will be examined.

ELIGIBILITY:
Inclusion criteria

* Female
* Proficiency in English
* Right-handed
* Between 19 and 60 years.
* Diagnosis of Anorexia Nervosa for participants in the clinical group.
* Body Mass Index between 18.5 and 25 kg/m² and no history of, or current, mood and anxiety disorders for participants in the healthy control group.

Exclusion criteria

* History of head trauma
* Hearing or visual impairment
* Neurological disease
* Claustrophobia
* Pregnancy
* Metal in the body which cannot be removed
* History of (or current) drugs and/or alcohol abuse
* Acute suicidality
* Psychotropic medication (other than antidepressants in the patient group).

Ages: 19 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2011-09; Primary Completion 2011-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Body mass index (body weight in kilograms divided by height in meters squared). | Approximately 3 months after the completion of the baseline questionnaires.
  Patients' weight and height are recorded.
Eating Disorder Examination Questionnaire (TOTAL subscale). | Approximately 3 months after the completion of the baseline questionnaires.
  Total score derived from 36 items. The items are rated using a Likert scale ranging from 0 to 6.
Visual analogue scale measuring anxiety symptoms. Participants are asked to answer the question "How anxious do you feel in this moment?" in response to viewing food pictures during a brain scan. | Approximately 3 months after the completion of the baseline questionnaires.
  Visual analogue scale ranging from 0 (not anxious at all) to 100 (extremely anxious).

SECONDARY OUTCOMES:
Likert scale measuring participants' confidence to challenge their eating disorder. | Approximately 3 months after the completion of the baseline questionnaires.
  Likert scale ranging from 0 (not confident at all) to 10 (very confident).

CONTACTS AND LOCATIONS:
Locations (1):
- Valentina Cardi, London, London, United Kingdom